CLINICAL TRIAL: NCT03439800
Title: Effects of Motor Imagery and Action Observation Training on Gait and Brain Activation Pattern of Individuals With Parkinson's Disease: Randomized Controlled Clinical Trial
Brief Title: Effects of Motor Imagery Training on Gait and Brain Activation Pattern of Individuals With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP-UFRN 2.057.658
Record Dates: First submitted 2017-11-15; First posted 2018-02-20 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Primary Parkinsonism; Rehabilitation; Kinematics; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental and Physical Practice (Experimental): Action observation: is defined as the observation of the motor action, in this study, through a video.
  Mental Practice: is defined as motor imagery training with the aim of improving the engine performance. Is the imagination of a motor action without its physical implementation.
  Physical Practice: is the execution of the motor action.
  Interventions: Other: Mental and Physical Practice
- Physical Practice (Active Comparator): Physical Practice: is the execution of the motor action.
  Interventions: Other: Physical Practice

INTERVENTIONS:
Other: Mental and Physical Practice — 1. Subjects will see a video of the typical gait and will attempt to analyze the sequence of the gait cycle.
  2. They will imagine themselves walking in the first-person perspective (kinesthetic) using the gait of the non-pathological pattern during 2 minutes.
  3. From the 1st to 4th session, the subjects will perform gait with corrections identified in previously in the video for 2 minutes.
  4. From 5th to 8th session: the subjects will do the protocol already described, however, the imagined gait will be in an environment with obstacles, also for 2 minutes. They will continue with the physical practice of the gait with obstacles.
  5. From 9th to final training session: both mental and physical practice of the dual task gait.
  Arms: Mental and Physical Practice
Other: Physical Practice — 1. Subjects will see a video about PD which does not mention physiotherapy treatments related to gait and they will explain their understanding about the theme.
  2. Then, the patients will make the physical gait protocol. Patients will be invited to perform the gait, in flat and firm ground with a length of 60 meters. The execution will be carried out for 10 minutes.
  3. From the 5th to 8th session, the subjects will do the physical practice of the gait with obstacles (which will be: going through 2 cones zigzag, going up and down 1 step, going through a narrow door, going up and down 1 ramp, going over 1 box of shoes, climbing a ramp, going down 1 step) for 2 minutes.
  4. From the 9th to the final training session, the subjects will do physical practice of the dual task gait.
  Arms: Physical Practice

SUMMARY:
INTRODUCTION: Mental practice (MP) and action observation (AO) are characterized as cognitive strategies that contribute to motor planning and learning in diverse populations. Individuals with Parkinson's Disease (PD) are recent targets, since, with disease progression, they need external strategies to aid in motor organization. However, there is still no evidence of the efficacy of MP and AO in the gait of PD. OBJECTIVES: To compare the effects of physical practice preceded by MP and AO on gait performance in individuals with Idiopathic PD (IPD). METHODS: A controlled, randomized, single-blind clinical trial with 66 individuals with IPD, aged between 50 and 75 years, without cognitive deficit and in the moderate phase of the disease will be performed. For the inclusion and characterization of the sample, the following instruments / equipment will be used: (1) Identification form (sociodemographic, clinical and anthropometric aspects); (2) Mini Mental State Examination and Montreal Cognitive Assessment (cognitive level); (3) Hoehn and Yahr Scale (level of physical disability); (4) Revised Movement Imagery Questionnaire (sharpness of the mental image); (5) Qualisys Motion Capture Systems® (gait kinematics); (6) Emotiv Epoc + (electroencephalographic activity); (7) Unified Parkinson's Disease Rating Scale - UPDRS (motor function and activities of daily living); (8) Timed Up and Go Test - TUG Test (mobility); and (9) Parkinson's Disease Questionnaire - PDQ-39 (quality of life).Participants included will be randomly assigned to two groups: experimental (n = 33), who will participate in MP + AO and physical gait practice; and control group (n = 33), who will participate only in the physical practice of gait. Both groups will be submitted to 12 training sessions (3x / week, for 4 weeks) and will be reevaluated 10 minutes, 7 days and 30 days after the last training session with respect to items (4), (5), (6) and (8) of the evaluation. Primary outcomes will be velocity, stride length and range of motion of the hip and the secondary ones will be sharpness of the mental image, electroencephalographic activity and performance in the TUG Test. The normality in the data distribution will be verified through the Shapiro-Wilk test. The "t" test and the Mann-Whitney test will be used to verify the homogeneity of the groups in the baseline. A repeated measures ANOVA will verify the interaction between the groups at the moments observed.

DETAILED DESCRIPTION:
No additional information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the report of a neurologist;
* Age between 50 and 75 years;
* In the moderate stage of the disease (between stages 2 and 3 of the Hoehn and Yahr Scale);
* Use of antiparkinsonian medication;
* Do not present cognitive deficits, according to the Mini Mental State Examination - MMSE. The cutoff point will be defined considering the individual's schooling (Illiterates: 18; With school instruction: 24);
* Ability to imagine motor acts in kinesthetic mode (according to the Revised Movement Imagery Questionnaire - MIQ-R). The cut-off point will be 20 for the kinesthetic modality, indicating that it is at least "a little easy to feel" the kinesthetically imagined movement;
* Have not undergone stereotaxic surgery.

Exclusion Criteria:

* Individuals with other associated neurological diseases;
* Individuals with musculoskeletal disorders, not related to the disease, but that impair gait;
* Individuals with hemodynamic instability before or during training;
* Individuals with uncorrected visual or auditory changes;
* Individuals who do not understand some stage of the training protocol.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Velocity | Change from Baseline Velocity at 1 day, 7 days and 30 days after training sessions
  Gait velocity in meters/second evaluated with Qualisys Motion Capture System

SECONDARY OUTCOMES:
Electroencephalographic activity | Change from Baseline Electroencephalographic activity at 1 day, 7 days and 30 days after training sessions
  Sharpness of the mental image evaluated by the Emotiv Epoc +
Mobility | Change from Baseline Mobility at 1 day, 7 days and 30 days after training sessions
  Performance in the Timed Up and Go Test
Stride length | change from Baseline Stride length at 1 day, 7 days and 30 days after training sessions
  Stride length during gait of the most affected lower evaluated with Qualisys Motion Capture System

CONTACTS AND LOCATIONS:
Locations (1):
- Lorenna Santiago, Parnamirim, Rio Grande Do Norte, Brazil

REFERENCES:
- [Derived] Nascimento IAPDS, Santiago LMM, de Souza AA, Pegado CL, Ribeiro TS, Lindquist ARR. Effects of motor imagery training of Parkinson's disease: a protocol for a randomized clinical trial. Trials. 2019 Nov 9;20(1):626. doi: 10.1186/s13063-019-3694-8. PMID 31706325